CLINICAL TRIAL: NCT00206232
Title: Novel Treatment for Diastolic Heart Failure in Women
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Karla Kurrelmeyer, MD, Baylor College of Medicine
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: H - 13988
Record Dates: First submitted 2005-09-12; First posted 2005-09-21 (Estimated); Last update posted 2013-02-18 (Estimated); Status verified 2013-02

CONDITIONS: Heart Failure
Keywords: Diastolic Heart Failure
MeSH Terms: conditions — Heart Failure; Heart Failure, Diastolic | interventions — Spironolactone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Spironolactone (Active Comparator): Randomized, double-blind, placebo controlled trial evaluating the safety and efficacy of spironolactone 25mg daily for 6 months.
  Interventions: Drug: Spironolactone
- Placebo (Placebo Comparator): Randomized, double-blind, placebo controlled trial evaluating the safety and efficacy of spironolactone 25mg daily for 6 months.
  Interventions: Drug: Spironolactone

INTERVENTIONS:
Drug: Spironolactone — Research subjects are randomized to placebo versus spironolactone 25mg daily and followed for 6 months.
  Other Names: Aldactone

SUMMARY:
The purpose of the study is to collect information about the potential benefit and safety of low dose spironolactone for a patient with diastolic heart failure (DHF) and to determine whether spironolactone can cause the patient's condition to improve.

DETAILED DESCRIPTION:
Subjects with diastolic heart failure defined based on clinical symptoms, echocardiography diastology parameters and brain natriuretic peptide level will be randomized in a 1:1 fashion to either placebo or spironolactone 25mg daily for 6 months. They will be assessed over this 6 month period for improvement in exercise capacity, clinical symptoms, echocardiography diastology parameters, and biomarkers specific for heart failure. Safety of spironolactone in this patient population will also be assessed by recording adverse events and following electrolytes, blood urea nitrogen, and creatinine levels.

ELIGIBILITY:
Inclusion Criteria:

* Women who are 18 years of age or older.
* Women with clinical heart failure for > 2 months.
* Women with left ventricular ejection fraction > 50% within 2 months of screening.
* Women with New York Heart Association class II or III heart failure symptoms.
* Brain Natriuretic Peptide > 62 pg/ml within 2 months of screening.
* Patient on angiotensin converting enzyme inhibitor or angiotensin receptor blocker therapy for at least 1 month.
* Blood Pressure no more than 150/95.
* Patient able to walk more than 50 meters at the time of enrollment.
* Signed informed consent.

Exclusion Criteria:

* Current treatment with spironolactone.
* Severe hepatic impairment.
* Creatinine > 2.5 mg/dl
* Potassium > 5.0 mEq/L
* Intolerance to spironolactone in the past.
* Significant valvular heart disease, pericardial disease, or severe chronic lung disease with cor pulmonale.
* Unstable angina or myocardial infarction within the past 4 weeks.
* Severe peripheral vascular disease or other physical conditions that would limit the walking distance.
* Pregnant or lactating females.
* Participation in any other drug trial within 30 days prior to randomization.
* Inability to provide informed consent.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2004-07; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Six minute walk distance | Baseline, then 3 and 6 months after randomization

SECONDARY OUTCOMES:
Echocardiography parameters of diastolic function | Baseline, then 3 and 6 months after randomization

OTHER OUTCOMES:
Procollagen peptides, troponin I, tumor necrosis factor alpha, Brain Natriuretic Peptide | Baseline then 3 and 6 months after randomization
Electrolytes, blood urea nitrogen, creatinine | Screening and enrollment then 10 days, 4 weeks, 11 weeks, 13 weeks, and 15 weeks after randomization
Quality of Life Questionaire | Baseline, then 3 and 6 months after randomization
New York Heart Association Classification | Baseline then 3 and 6 months after randomization
Number of participants with adverse events | From randomization until trial completion at 6 months.

CONTACTS AND LOCATIONS:
Overall Officials: Karla M Kurrelmeyer, MD, Principal Investigator — Baylor College of Medicine
Locations (1):
- Baylor College of Medicine Heart Clinic, Houston, Texas, United States

REFERENCES:
- [Derived] Kurrelmeyer KM, Ashton Y, Xu J, Nagueh SF, Torre-Amione G, Deswal A. Effects of spironolactone treatment in elderly women with heart failure and preserved left ventricular ejection fraction. J Card Fail. 2014 Aug;20(8):560-8. doi: 10.1016/j.cardfail.2014.05.010. Epub 2014 Jun 4. PMID 24905296